CLINICAL TRIAL: NCT07385781
Title: Psychosomatic Symptoms in Patients With Myofascial Pain and Temporomandibular Joint Dysfunction- A Case Control Study
Brief Title: Psychosomatic Symptoms in Patients With Myofascial Pain and Temporomandibular Joint Dysfunction
Acronym: Psychosomatic
Status: Not yet recruiting | Type: Observational
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Dr Rida Zulfiqar, Registrar, Bahria University
Other Study IDs: 17/2023; bahria university (Other: bahria university)
Record Dates: First submitted 2025-12-11; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Psychosomatic Symptoms; Temporomandibular Disorder (TMD)
Keywords: Anxiety; Depression; myofascial facial pain; Perceived stress; Somatization
MeSH Terms: conditions — Temporomandibular Joint Disorders; Anxiety Disorders; Depression | interventions — Receptors, Calcium-Sensing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: A total of 300 participants aged between 20 and 60 years were recruited using survivor sampling, consisting of 150 patients with a confirmed diagnosis of myofascial pain and temporomandibular joint dysfunction (TMD) and 150 age- and gender-matched healthy controls
  Interventions: Other: Casr
- Control: A total of 300 participants aged between 20 and 60 years were recruited using survivor sampling, consisting of 150 patients with a confirmed diagnosis of myofascial pain and temporomandibular joint dysfunction (TMD) and 150 age- and gender-matched healthy controls
  Interventions: Other: Casr

INTERVENTIONS:
Other: Casr — case study participants

SUMMARY:
Background: Temporomandibular joint disorder poses an intricate etiology. Biomechanical, neuromuscular and psychosocial factors may contribute to the disorder among which psychological and psychosocial disturbances have shown strong direct or indirect contribution to the disease especially when the pain is of muscular origin.

Objective: To investigate psychosomatic symptoms among patients with myofascial pain & temporomandibular joint dysfunction from 20 to 60 years of age.

Methodology: This multicentre case-control study included 300 participants aged 20-60 years, comprising 150 clinically diagnosed TMD cases and 150 matched healthy controls. Clinical evaluation was performed using the Research Diagnostic Criteria for TMD (RDC/TMD Axis I), assessing joint mobility, muscle tenderness, and mandibular function. Psychosomatic symptom burden was evaluated using the Symptom Checklist-27 (SCL-27), covering six domains: depressive, dysthymic, vegetative, agoraphobic, social phobia, and mistrust symptoms. Independent t-tests and chi-square analyses were used to compare group differences, with significance set at p < 0.05.

DETAILED DESCRIPTION:
Introduction Temporomandibular disorders (TMDs) are defined as the group of musculoskeletal and neuromuscular conditions that involves temporomandibular joint (TMJ), masticatory muscles, and their associated structures (1). Clinically, TMDs are characterized by jaw pain, mandibular movement limitation, joint sounds, and often referred pain in the head, neck, or shoulders region (2). The myofascial pain, a subtype of TMD, is most prevalent condition and it accounts for approximately 50% of all TMD cases in clinical settings (3). Although it's a prevalent condition, but its complex aetiology makes it difficult to diagnose (4).

Recent advances in dentistry have categorised TMD to a biopsychosocial disorder rather than pure biomechanical issue, implicating emotional distress, behavioural patterns, and environmental stressors in both the onset and progression of symptoms (5). Psychological comorbidities such as depression, anxiety, and somatization are frequently reported in individuals with TMD (6). These symptoms have a tendency to influence perception of pain, coping strategies, and treatment adherence which results in complicating the clinical outcomes. The recognition of these non-structural contributors is now added in diagnostic systems such as the Diagnostic Criteria for TMD (DC/TMD), which includes both Axis I (physical diagnosis) and Axis II (psychosocial status and pain-related disability) assessments (7).

Myofascial pain syndrome (MPS) is defined by the presence of trigger points and referred pain patterns in the masticatory muscles. Its prevalence ranging from 9% to 21% in the general population, however it is higher among individuals who experience psychological stress or mood disorders (8). Several studies have demonstrated that stress-related activities such as bruxism, jaw clenching, and tongue thrusting act as mediators between emotional dysregulation and muscular overactivity, thus aggravating MPS and contributing to the chronicity of pain (9). Moreover, the chronic nature of MPS often leads to central sensitization, amplifying pain signals and establishing a vicious cycle of pain and distress (9).

Psychosomatic symptoms are the physical symptoms that arise or exacerbated by emotional factors. Psychosomatic manifestations such as headaches, jaw discomfort, tinnitus, and even dizziness may not be explained entirely by anatomical or mechanical abnormalities in TMDS. The Symptom Checklist-27 (SCL-27) is a validated instrument for screening depressive, anxiety-related, vegetative, and social phobia symptoms. This tool is used in several studies to assess psychological distress in orofacial pain disorders (10).

While a growing body of literature from Western research has reported the link between psychosocial factors and TMD, however, there remains a notable gap in evidence from South Asian populations, where stigma associated with mental health, cultural issues, and limited access to psychological services may significantly affect clinical presentations. In Pakistan oral health care delivery is primarily dentist-centred and biomedical in focus. The integration of psychosocial evaluation into TMD management remains largely unexplored. Moreover, there is a growing consensus among global pain specialists that a multidisciplinary and integrative treatment approach that involves mental health professionals yields superior outcomes for TMD patients with comorbid psychosomatic disturbances. Therefore, the current study aims to investigate psychosomatic symptoms in patients diagnosed with myofascial pain and temporomandibular joint dysfunction Materials and Methods The study protocol was approved by the Institutional Ethics Committee. Participants were assured of the confidentiality of their responses, and the data were anonymized before analysis. No financial or therapeutic incentives were provided. This study was designed as a multicentre, matched case-control study conducted at public and private dental colleges in Karachi, Pakistan, between March 2022 and December 2022. The study adhered to the principles outlined in the Declaration of Helsinki (2013) (11).

A total of 300 participants aged between 20 and 60 years were recruited using survivor sampling, consisting of 150 patients with a confirmed diagnosis of myofascial pain and temporomandibular joint dysfunction (TMD) and 150 age- and gender-matched healthy controls. All participants were briefed about the study objectives, and written informed consent was obtained prior to data collection. The inclusion criteria for case group participants included diagnosed patients with myofascial pain and TMD for at least six months based on Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD), Axis I, age between 20 and 60 years, literate and able to comprehend the questionnaire and with no prior psychological treatment for pain. In control group, the healthy individuals without symptoms of myofascial pain or TMD, matched for age and gender with cases, no known psychiatric illness or chronic pain condition and with no clinical signs of TMD upon examination were included. The individuals were excluded if the age was <20 or >60 years, low literacy (less than five years of formal education), history of major psychiatric or neurological disorders, diagnosed joint pathologies (e.g., arthritis, disc displacement with reduction), history of migraine or facial trauma, drug dependency and pregnancy or current use of psychotropic medication.

Sample size was calculated using OpenEpi® version 3.01, based on an expected effect size of 0.4 (moderate), with a power of 80% and a 5% level of significance. The minimum required sample size was 134 participants per group. To account for potential dropouts and non-responses, a total of 150 subjects were included in each group.

Clinical Examination Protocol All clinical assessments were conducted by calibrated examiners trained in the use of the RDC/TMD protocol to ensure standardization and inter-rater reliability. The clinical examination included palpation of masticatory and cervical muscles using 2 kg/cm² of pressure for 5 seconds, based on RDC/TMD muscle examination guidelines. The muscles examined were masseter, temporalis (anterior and posterior), medial and lateral pterygoid, sternocleidomastoid, trapezius, and occipital insertion points. Mandibular range of motion, including maximum mouth opening (in mm), lateral excursions (left and right) and protrusive movements were recorded. Pain responses were graded from 0 to 3 i-e., 0: No pain, 1: Discomfort, 2: Moderate pain, and 3: Severe pain. TMJ function was evaluated through observation of opening patterns (deviation/deflection), presence of joint sounds (clicking, crepitus), and palpation of the joint during mandibular movements.

The Symptom Checklist-27 (SCL-27) was used to assess psychosomatic symptoms across six domains i-e., depressive symptoms, dysthymic symptoms, vegetative symptoms, agoraphobic symptoms, social phobia and mistrust and suspiciousness. Each item was rated on a 5-point Likert scale ranging from "strongly disagree" (1) to "strongly agree" (5). The SCL-27 has been previously validated in clinical populations and exhibits high internal consistency (Cronbach's alpha > 0.85 for most subscales). Participants completed the SCL-27 under the supervision of the research team to ensure completeness and accuracy. Data with missing values >10% per scale were excluded from analysis.

ELIGIBILITY:
Inclusion Criteria:

diagnosed patients with myofascial pain and TMD for at least six months based on Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD), Axis I, age between 20 and 60 years, literate and able to comprehend the questionnaire no prior psychological treatment for pain.

Exclusion Criteria:

age <20 or >60 years, low literacy (less than five years of formal education), history of major psychiatric or neurological disorders, diagnosed joint pathologies (e.g., arthritis, disc displacement with reduction), history of migraine or facial trauma, drug dependency and pregnancy or current use of psychotropic medication.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Temporomandibular joint dysfunction patient
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Psychosomatic symptom burden | 2 months
  Psychosomatic symptom burden is defined as the overall severity and frequency of physical symptoms that are influenced or maintained by psychological factors. It will be assessed using a validated self-report questionnaire that captures multiple somatic symptom domains (e.g., pain, gastrointestinal, cardiovascular, and fatigue-related symptoms). Higher scores indicate a greater psychosomatic symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Rida Zulfiqar, Principal Investigator — Bahria University
Locations (1):
- Bahria University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: jan 2026-Dec2026

REFERENCES:
- [Result] 1. Szarejko KD, Gołębiewska M, Lukomska-Szymanska M, Kuć J. Stress experience, depression and neck disability in patients with temporomandibular disorder-myofascial pain with referral. Journal of Clinical Medicine. 2023;12(5):1988. 2. Kuć J, Szarejko KD, Maciejczyk M, Dymicka-Piekarska V, Żendzian-Piotrowska M, Zalewska A. Oxidative imbalance as a co-player in jaw functional limitations and biopsychosocial profile in patients with temporomandibular disorder-Myofascial pain with referral. Frontiers in Neurology. 2025;15:1509845. 3. Gomes AKP, Ximenes TA, Fonseca APR, de Barros Silva PG, Magalhães IA, da Silva Rodrigues AK, et al. Relationship between temporomandibular joint dysfunctions and psychosomatic factors. Revista Eletrônica Acervo Saúde. 2024;24(5):e16019-e. 4. Syroishko M, Kostiuk T. Dysfunction of the temporomandibular joints associated with post-traumatic stress disorders in patients. Reports of Vinnytsia National Medical University. 2023;27(2):253-7. 5. Matos M, Thumati P, Sutter B, Ruiz-Velasco G, Goldberg J, Booth J, et al. Are Temporomandibular Disorders Really Somatic Symptom Disorders? Part II-Joint Vibration Analysis of the Temporomandibular Joint. Advanced Dental Technologies & Techniques. 2021. 6. Patil DJ, Dheer DS, Puri G, Konidena A, Dixit A, Gupta R. Psychological appraisal in temporomandibular disorders: A cross-sectional study. Indian Journal of pain. 2016;30(1):13-8. 7. Canales GDLT, Guarda-Nardini L, Rizzatti-Barbosa CM, Conti PCR, Manfredini D. Distribution of depression, somatization and pain-related impairment in patients with chronic temporomandibular disorders. Journal of Applied Oral Science. 2019;27:e20180210. 8. Urits I, Charipova K, Gress K, Schaaf AL, Gupta S, Kiernan HC, et al. Treatment and management of myofascial pain syndrome. Best Practice & Research Clinical Anaesthesiology. 2020;34(3):427-48. 9. Cao Q-W, Peng B-G, Wang L, Huang Y-Q, Jia D-L, Jiang H, et al. Expert consensus on the diagnosis and treatment of myofascial pai
- [Result] Szarejko KD, Golebiewska M, Lukomska-Szymanska M, Kuc J. Stress Experience, Depression and Neck Disability in Patients with Temporomandibular Disorder-Myofascial Pain with Referral. J Clin Med. 2023 Mar 2;12(5):1988. doi: 10.3390/jcm12051988. PMID 36902775